CLINICAL TRIAL: NCT06882954
Title: The Management of Asymptomatic Carotid Stenosis: Monocentric Experience
Brief Title: The Management of Asymptomatic Carotid Stenosis
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Associate Professor of Vascular Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2691
Record Dates: First submitted 2023-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Carotid Artery Diseases; Carotid Stenosis
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carotid stenosis are asymptomatic if no hemispheric or retinal symptoms have appeared in the 6 months preceding the discovery of the stenosis. Asymptomatic carotid stenosis (ACS) accounts for about ¾ of all carotid lesions. The goal of treating carotid stenosis is to prevent a stroke. While carotid surgery is recommended in the elderly patients in cases of symptomatic carotid stenosis, that of ACS in patients over 75 years old, even when tight, remains subject to many controversies. Indeed, the debate, concerning the benefit to be expected from a surgical procedure or a possible angioplasty procedure, is not yet closed. The aim of our study, through a retrospective evaluation of the results of all consecutive carotid endarterectomy (CEA) and stenting in the participating center.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic carotid stenosis
* Patient with degree of carotid stenosis greater than 80% measured by the maximum systolic velocity at the site of the stenosis which must have been greater than 250 cm/s
* Ultrasound characteristics of a possibly unstable plaque

Exclusion Criteria:

* Symptomatic carotid artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with significant internal carotid artery stenosis referred to the Unit of Vascular Surgery of Fondazione Policlinico Gemelli IRCCS Rome for carotid artery endoarterectomy and stenting
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke rate | Through study completion, an average of 1 year
  Rate of stroke after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No